CLINICAL TRIAL: NCT06654778
Title: Ultrasound Evaluation of Different Preventive Measures of Post Operative Lung Atelectasis After Upper Abdominal Surgeries: Ventilation and Fluid Measures
Brief Title: Ultrasound Evaluation of Preventive Measures for Postoperative Lung Atelectasis After Surgery
Acronym: LUS/PEEP/RM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hamed Mohamed Wally Allah, Assistant lecturer in Anesthesia, Intensive Care and pain management department, Faculty of Medicine, Al-Azhar University (Assiut), Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AZAST/MD/209/MARCH/2024
Record Dates: First submitted 2024-10-20; First posted 2024-10-23 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Atelectasis, Postoperative
Keywords: lung ultrasound; lung Atelectasis; Atelectasis; Pulmonary Atelectasis; pressure controlled ventilation - volume guarantee (PCV- VG); positive end-expiratory pressure (PEEP); lung recruitment maneuver; restrictive fluid strategies
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: The patients will be assigned into three equal groups of 20 patients each:
  1. Group I: PEEP of 8 cm H2O and fluid management: 500 ml + 4 mL/kg/hour Ringer's lactate
  2. Group II: PEEP/RM group, addition of RM (30 cm H2O for 30 s)
  3. Group III: PEEP/RM group and restricted fluid management 3 mL/kg/hour Ringer's lactate
  A total sample size of 60 patients will be involved.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: PEEP (Experimental): Patients will be ventilated with PEEP of 8 cm H2O and fluid management: 500 ml of Ringer's lactate in the recovery room before surgery and Ringer's lactate at a rate of 4 mL/kg/hour from the beginning to the end of the surgery.
  Interventions: Other: PEEP
- Group II: PEEP/RM (Experimental): Patients will be ventilated with PEEP of 8 cm H2O, and then RM (30 cm H2O for 30 s) will be applied immediately after the second LUS examination and repeated every 30 minutes till emergence and fluid management: 500 ml of Ringer's lactate in recovery room before surgery and Ringer's lactate at a rate of 4 mL/kg/hour from the beginning to the end of the surgery
  Interventions: Other: PEEP/RM
- Group III: PEEP/RM/RF (Experimental): Patients will be ventilated with PEEP of 8 cm H2O, and then RM (30 cm H2O for 30 s) will be applied immediately after the second LUS examination and repeated every 30 minutes till emergence and restrictive fluid management (RF). Ringer's lactate at a rate of 3 mL/kg/hour from the beginning to the end of the surgery
  Interventions: Other: PEEP/RM/RF

INTERVENTIONS:
Other: PEEP — Patients will be ventilated with PEEP of 8 cm H2O and fluid management: 500 ml of Ringer's lactate in the recovery room before surgery and Ringer's lactate at a rate of 4 mL/kg/hour from the beginning to the end of the surgery.
  Arms: Group I: PEEP
Other: PEEP/RM — Patients will be ventilated with PEEP of 8 cm H2O, and then RM (30 cm H2O for 30 s) will be applied immediately after the second LUS examination and repeated every 30 minutes till emergence and fluid management: 500 ml of Ringer's lactate in recovery room before surgery and Ringer's lactate at a rate of 4 mL/kg/hour from the beginning to the end of the surgery
  Arms: Group II: PEEP/RM
Other: PEEP/RM/RF — Patients will be ventilated with PEEP of 8 cm H2O, and then RM (30 cm H2O for 30 s) will be applied immediately after the second LUS examination and repeated every 30 minutes till emergence and restrictive fluid management (RF). Ringer's lactate at a rate of 3 mL/kg/hour from the beginning to the end of the surgery
  Arms: Group III: PEEP/RM/RF

SUMMARY:
the aim of this prospective randomized blinded clinical study will be to assess the ultrasound evaluation of different preventive measures of post operative lung atelectasis in abdominal surgeries; these measures include ventilation and fluid measures

DETAILED DESCRIPTION:
ultrasound evaluation for application of different preventive measures of post operative lung atelectasis, including positive end-expiratory pressure, lung recruitment maneuvers, and restrictive fluid management.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II, of either gender.
* BMI < 40
* Age 30-60 years
* scheduled for elective abdominal surgeries

Exclusion Criteria:

* Patient refusal
* American Society of Anesthesiologists (ASA) physical status classification system more than II
* BMI > 40 .
* Psychiatric disorders
* History of chest disorders such as asthma and obstructive pulmonary disease (COPD).
* History of Previous Thoracic Procedures.
* Pregnancy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-08 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Lung ultrasound assessment of postoperative pulmonary atelectasis at the end of surgery | at the end of surgery before emergence from GA.
  Lung ultrasound assessment of postoperative pulmonary atelectasis at the end of surgery.
  The Lung Ultrasound Score (LUS): the key points based on ultrasound findings:
  I. 0 points: (N) Normal aeration (presence of lung sliding with A-lines or <2 separate B-lines).
  II. 1 point: (B1) Moderate loss of lung aeration (≥3 well-defined B lines). III. 2 points: (B2) Severe loss of lung aeration (coalescing B-lines). IV. 3 points: (C) Complete loss of lung aeration (pulmonary consolidations). Total Score: points will be distributed according to the worst ultrasound pattern observed: N = 0, B1 lines = 1, B2 lines = 2, C = 3. The LUS score ranging between 0 and 36 was calculated as the sum of points.

SECONDARY OUTCOMES:
Lung ultrasound assessment | before induction of general anesthesia
  Lung ultrasound assessment of atelectasis
Lung ultrasound assessment | 5 minutes post induction of general anesthesia
  Lung ultrasound assessment of atelectasis
Lung ultrasound assessment | 15 minutes after patients arrive to PACU
  Lung ultrasound assessment of atelectasis
Lung ultrasound assessment | 60 minutes after patients arrive to PACU
  Lung ultrasound assessment of atelectasis
arterial blood gases | 5 minutes post induction of general anesthesia
  Pao2, spo2, paco2, pao2/fio2
arterial blood gases | before emergence from general anesthesia
  Pao2, spo2, paco2, pao2/fio2
arterial blood gases | 15 minutes after patients arrive to PACU
  Pao2, spo2, paco2, pao2/fio2

CONTACTS AND LOCATIONS:
Overall Officials: Hamed M Wally Allah, Principal Investigator — Al-Azhar University
Locations (1):
- Al-Azhar university, Asyut, Egypt